CLINICAL TRIAL: NCT07315191
Title: The Randomized Controlled Trial of Finerenone Therapy for Pediatric Hennoch Scholein Nephritis With Mild Proteinuria
Brief Title: Finerenone Therapy for Pediatric HSPN With Mild Proteinuria
Acronym: FICHSPN
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Capital Institute of Pediatrics, China (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BRWEP2024W102100109
Record Dates: First submitted 2025-12-18; First posted 2026-01-02 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Henoch Schönlein Purpura Nephritis
MeSH Terms: interventions — Angiotensin-Converting Enzyme Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Finerenone group (Experimental)
  Interventions: Drug: ACEI / ARB+finerenone
- Control group (Active Comparator)
  Interventions: Drug: ACEI/ARB

INTERVENTIONS:
Drug: ACEI / ARB+finerenone — In the finerenone group, finerenone was administered orally on the basis of combined oral ACEI/ARB, with the dose calculated based on body surface area, once a day for 3 months.
  Arms: Finerenone group
Drug: ACEI/ARB — The control group was only given oral ACEI/ARB for 3 months.
  Arms: Control group

SUMMARY:
Henoch-Schönlein purpura nephritis (HSPN) is the most common secondary glomerular disease in children. About 40% of HSPN cases are accompanied by mild proteinuria, and some of them progress to end-stage renal disease. Currently, the treatment for children with mild proteinuria HSPN mainly involves ACEI/ARB, but long-term use of these drugs can lead to an increase in aldosterone levels, affecting therapeutic efficacy. Finerenone can improve vascular endothelial cell dysfunction and renal tissue inflammation and fibrosis, and reduce urinary protein in patients with glomerular diseases. This study intends to conduct an exploratory randomized controlled clinical trial of finerenone in children with HSPN accompanied by a small amount of proteinuria to evaluate the efficacy and safety of finerenone treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Children of HSPN meet the following conditions① Age > 3 years old and < 18 years old;
2. 24-hour urine protein quantification >= 8mg/h/M2 body surface area (or >= 300mg/d), and < 20mg/h/M2 body surface area (< 1000mg/d);

3: 3. Sign the informed consent form.

Exclusion Criteria:

1. Abnormal renal function: eGFR < 90 ml/min/1.73m^2 body surface area;
2. Renal pathological grade >= IV;
3. Application of glucocorticoids and/or immunosuppressants within 2 weeks;
4. Recent applications involving high-dose glucocorticoids administered for a duration exceeding two weeks.;
5. Liver transaminase > 2 times the upper limit of normal;
6. Severe cardiac insufficiency;
7. Simultaneous use of CYPA4 inhibitors;-

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 116 (Estimated)
Dates: Start 2025-06-13 (Actual); Primary Completion 2027-10-31 (Estimated); Study Completion 2028-04-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of Subjects with a Reduction in 24-Hour Urinary Protein Excretion ≥30% from Baseline | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Capital Center for Children's Health,Capital Medical University, Beijing, Beijing Municipality, China